CLINICAL TRIAL: NCT03646851
Title: Impact of Aspergillus on Chronic Obstructive Pulmonary Disease Evolution
Brief Title: Aspergillus and Chronic Obstructive Pulmonary Disease Evolution
Acronym: AspergBPCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PI2017_843_0024
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD (Experimental): COPD patients GOLD stage III and IV
  Interventions: Diagnostic Test: Questionnaries

INTERVENTIONS:
Diagnostic Test: Questionnaries — patients will have to do a sputum and to complete some questionnaries

SUMMARY:
This is a prospective multicenter cohort study which includes all consecutive COPD patients who come for a visit in one the participating pneumologist. They will have to do a sputum and to complete some questionnaries. Questionnaries will be redone by phone after 1 and 3 months and during the visit after 6 months. We will correlate aspergillus presence in sputum with quality of life (QoL), and COPD symptoms evaluated by questionnaires.

DETAILED DESCRIPTION:
Aspergillosis disease is a growing problem. These diseases are not yet uncommon in chronic obstructive pulmonary disease patients. (COPD).

Aspergillosis disease are very difficult to be diagnosed or treated. Isolation of aspergillus in sputum of patients is not always responsible of a real disease. Need of treatment is discussed. That is why, we will conduct a prospective cohort study to evaluate aspergillus rate in respiratory samples of COPD patients (GOLD stage III or IV)

ELIGIBILITY:
Inclusion Criteria:

* COPD patients GOLD stage III and IV

Exclusion Criteria:

* Cystic fibrosis
* Pulmonary fibrosis
* hematological malignancy
* known aspergilloma
* allergic bronchopulmonary aspergillosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
presence of aspergillus in sputum or respiratory samples | one year before inclusion
  sputum examination

SECONDARY OUTCOMES:
Dyspnea with MMRC score | day of inclusion
  Pulmonary function testing

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CH Abbeville, Abbeville
  - CHU Amiens-Picardie, Amiens
  - Clinique de l'Europe, Amiens
  - CHU St Quentin, Saint-Quentin

IPD SHARING:
Plan to Share IPD: Undecided